CLINICAL TRIAL: NCT05333224
Title: Effectiveness of Telerehabilitation-Based Family-Centered Goal-Directed Physiotherapy Approach in High Risk of Infants
Brief Title: Effectiveness of Telerehabilitation in High Risk of Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 09.2021.853
Record Dates: First submitted 2022-01-13; First posted 2022-04-18 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2023-09

CONDITIONS: Early Intervention
Keywords: Risky Baby; Telerehabilitation; Family-centered approach; Early Intervention; Goal-directed physiotherapy
MeSH Terms: interventions — Telerehabilitation; Home Care Services, Hospital-Based

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation (Experimental): Mothers attended monthly exercise sessions at the hospital and engaged in home exercises for 45 minutes, twice weekly. They communicated their progress via messaging. Moreover, a 45-minute physiotherapy session was held weekly through live video conferencing, during which the physiotherapist guided and observed the mother while she interacted with a simulated infant model.
  Interventions: Other: Telerehabilitation
- Home-based (Other): Mothers underwent monthly exercise sessions at the hospital and engaged in home exercises lasting 45 minutes, thrice weekly. They documented their exercise routines on a weekly chart and discussed them with the physiotherapist during their monthly hospital appointments.
  Interventions: Other: Home-based

INTERVENTIONS:
Other: Telerehabilitation — Family-centered, goal-oriented early physiotherapy approaches will be applied.
  Arms: Telerehabilitation
Other: Home-based — Family-centered, goal-oriented early physiotherapy approaches will be applied.
  Arms: Home-based

SUMMARY:
While the mortality rate in preterm births has decreased thanks to recent developments in the field of medicine, disability risk factors increase for premature babies. Premature birth, low birth weight, and all accompanying problems in this process reveal the concept of the risky baby. Early intervention is very important for these babies who are at risk for neurodevelopmental problems. Although early intervention is a general concept, the subject the investigators focus on is early physiotherapy approaches. Early physiotherapy approaches include many methods. However, recently, family-centered approaches have been emphasized and studies have been carried out on this issue; Likewise, the goal-oriented therapy approach, which is a treatment with a high level of evidence, is also being investigated. Telerehabilitation, on the other hand, has become a method that is frequently used with the increase in the use of technological methods. The effectiveness of family-centered, goal-oriented physiotherapy approaches is known in previous studies on this subject; There are studies conducted on a remotely monitored portable intelligent system created for telerehabilitation, but no studies have been found in which telerehabilitation has been applied using the real-time video conferencing method.

DETAILED DESCRIPTION:
Babies in whom negative biological and environmental factors cause neuromotor developmental problems are defined as "risk babies". Risky babies are classified differently. This classification; may be according to gestational age, birth weight, and pathophysiological problems. Especially, premature babies born at 32 weeks and under 1500 g, babies with periventricular leukomalacia, hypoxic-ischemic encephalopathy, intraventricular hemorrhage, and intrauterine growth retardation are in the high-risk group.

The mortality rate in risky babies has decreased considerably in recent years, but with this decrease, neurodevelopmental disorders including motor problems, incoordination, cognitive impairment, attention problems, or developmental problems are seen in these babies who live prematurely, and the risk of Cerebral Palsy (CP) occurs. CP is the common name of a group of non-progressive permanent disorders that primarily lead to impairment in movement and posture development and activity limitation, and that can also be seen in addition to sensory and cognitive problems, due to permanent damage to the developing brain. The primary condition for early intervention is to identify babies who may have CP. Early detection may be beneficial for the initiation of early intervention in the period when neuroplasticity is high. Based on neuroplasticity knowledge, it is thought that it will be beneficial for risky babies during development, and it may be possible to prevent neurodevelopmental problems and permanent disabilities, with early intervention and protective approaches. In general, the early intervention approach includes supporting the development of babies who are at risk for developmental delay or disability by providing the necessary support, treatment, and training, starting from the neonatal period and up to 24 months. Early intervention methods have many components and require a multidisciplinary approach. Methods can focus on different approaches according to the determined goals. Physiotherapy and rehabilitation approaches are of great importance in supporting the development and improving functional outcomes in early intervention. It is aimed to provide normal sensory input and gain normal functional movements by using the rapid learning ability originating from brain plasticity, and to reach the most independent level that the child can reach in terms of physical, cognitive, and psychosocial aspects within the anatomical and physiological deficiencies and environmental limitations. There are many early physiotherapy and rehabilitation approaches that focus on motor development and normalization.

Goal-oriented therapy; is known as an approach that facilitates the participation and adaptation of infants and children with motor developmental delay to daily life activities. Goal-oriented neuromotor therapy approach; It is a set of movements organized around a functional goal and the environment enables the movement to occur. Studies on rehabilitation have recently focused on treatment approaches that focus on functionality in accordance with the "Activity and Participation" area of ICF. It is known that babies also have levels of functionality that enable them to participate in activities of daily living. In a study in which goal-oriented neuromotor therapy was applied in early rehabilitation applications, it was stated that this approach could be applied by both the physiotherapist and the family under the control of the physiotherapist. Family-centered physiotherapy applications have come to the fore in recent years, it is the treatment approach that focuses on the environment and what the child can do and practiced by family. Motor reactions are activated by providing normal sensory input. Telerehabilitation is the delivery of rehabilitation services by computer-based technologies and communication tools by rehabilitation specialists. It is an emerging method that provides rehabilitation services by reducing time, distance, and cost barriers and using technological tools.

Although the importance of early physiotherapy approaches is known today, when the literature is examined, it is seen that the number of studies is insufficient and a consensus has not yet been reached on which therapy approach is more successful. No study has been found in which family education of risky infants was followed up with telerehabilitation before.

ELIGIBILITY:
Inclusion Criteria:

* Babies born before <37 weeks of gestation and treated in the neonatal intensive care unit
* Infants with neurologic abnormalities (muscle hypertonia, hypotonia, hyperarousal, and abnormal general movements or cranial ultrasound abnormalities) at moderate to high risk of cerebral palsy
* Babies referred to physiotherapy due to motor developmental delay and neurological dysfunction
* Babies whose age range is between 0-12 months (corrected age will be calculated for premature babies)
* Being diagnosed as a neurologically and developmentally risky baby
* Babies who have completed their medical treatment and are not in neonatal intensive care
* Babies of families who agreed to participate in the study and approved the informed consent form.

Exclusion Criteria:

* Babies with congenital cyanotic heart problems or cystic fibrosis
* Babies with genetic disease or congenital anomaly
* Infants on ventilator
* Babies of families who do not accept to work
* Babies of families who cannot come to the control
* Families that cannot be contacted every week
* Babies going to a special education and rehabilitation center

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ayca Evkaya Acar, MSc, Principal Investigator — Istanbul Medeniyet University; Esra Pehlivan, Assoc. Prof., Study Director — Saglik Bilimleri University; Evrim Karadag Saygi, Prof., Principal Investigator — Marmara University
Locations (1):
- Marmara University Pendik Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asztalos EV, Church PT, Riley P, Fajardo C, Shah PS; Canadian Neonatal Network and Canadian Neonatal Follow-up Network Investigators. Association between Primary Caregiver Education and Cognitive and Language Development of Preterm Neonates. Am J Perinatol. 2017 Mar;34(4):364-371. doi: 10.1055/s-0036-1592080. Epub 2016 Aug 29. PMID 27571484
- [Background] Beaino G, Khoshnood B, Kaminski M, Marret S, Pierrat V, Vieux R, Thiriez G, Matis J, Picaud JC, Roze JC, Alberge C, Larroque B, Breart G, Ancel PY; EPIPAGE Study Group. Predictors of the risk of cognitive deficiency in very preterm infants: the EPIPAGE prospective cohort. Acta Paediatr. 2011 Mar;100(3):370-8. doi: 10.1111/j.1651-2227.2010.02064.x. Epub 2011 Jan 17. PMID 21241364
- [Background] Cameron EC, Maehle V, Reid J. The effects of an early physical therapy intervention for very preterm, very low birth weight infants: a randomized controlled clinical trial. Pediatr Phys Ther. 2005 Summer;17(2):107-19. doi: 10.1097/01.pep.0000163073.50852.58. PMID 16357661
- [Background] Draper ES, Zeitlin J, Manktelow BN, Piedvache A, Cuttini M, Edstedt Bonamy AK, Maier R, Koopman-Esseboom C, Gadzinowski J, Boerch K, van Reempts P, Varendi H, Johnson SJ; EPICE group. EPICE cohort: two-year neurodevelopmental outcomes after very preterm birth. Arch Dis Child Fetal Neonatal Ed. 2020 Jul;105(4):350-356. doi: 10.1136/archdischild-2019-317418. Epub 2019 Nov 5. PMID 31690558
- [Background] Guellec I, Lapillonne A, Renolleau S, Charlaluk ML, Roze JC, Marret S, Vieux R, Monique K, Ancel PY; EPIPAGE Study Group. Neurologic outcomes at school age in very preterm infants born with severe or mild growth restriction. Pediatrics. 2011 Apr;127(4):e883-91. doi: 10.1542/peds.2010-2442. Epub 2011 Mar 7. PMID 21382951

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Informed consent was obtained, and 26 infants and 26 mothers who presented to the high-risk infant clinic at Marmara University Hospital between 2022 and 2023 were included in the study.
Pre-assignment Details: After obtaining informed consent from the parents, 26 infants and 26 mothers were randomized into groups and assessments were conducted. However, a total of 2 infants and 2 mothers, one from each group, did not attend the follow-up evaluations at the hospital one month later, and thus were excluded from the study.
Groups:
- Telerehabilitation: A telerehabilitation-based exercise group where the therapist coaches the family, performs one-on-one exercises with families with a doll in his hand, and can perform the necessary interventions such as promoting good practices and preventing bad practices, and the other 2 days where the families show their exercises by sending videos to the therapist, and again provide the therapist's intervention and follow-up via videos.
  Telerehabilitation: Family-centered, goal-oriented early physiotherapy approaches will be applied.
- Control (Home-based Group): The Home-based group that will be given exercise training at the beginning of treatment and at 4., 8., and 12. week.
  Control: Family-centered, goal-oriented early physiotherapy approaches will be applied.
Period: Overall Study - Infants
Arm/Group | Telerehabilitation | Control (Home-based Group)
Started | 13 | 13
Completed | 12 | 12
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Period: Overall Study - Mothers
Arm/Group | Telerehabilitation | Control (Home-based Group)
Started | 13 | 13
Completed | 12 | 12
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Population: Risky babies with corrected ages ranging from 0-12 months and their mothers who applied to Risky Baby Polyclinic and babies who met the inclusion criteria.
Groups:
- Telerehabilitation - Infants: A telerehabilitation-based exercise group where the therapist coaches the family, performs one-on-one exercises with families with a doll in his hand, and can perform the necessary interventions such as promoting good practices and preventing bad practices, and the other 2 days where the families show their exercises by sending videos to the therapist, and again provide the therapist's intervention and follow-up via videos
  Telerehabilitation: Family-centered, goal-oriented early physiotherapy approaches will be applied.
- Home-based - Infants: The home-based group that will be given exercise training at the beginning of treatment and at 4., 8., and 12. week.
  Home-based: Family-centered, goal-oriented early physiotherapy approaches will be applied.
- Telerehabilitation -Mothers: Mothers exercising in the telerehabilitation group
- Home-based - Mothers: Mothers exercising in the control group
- Total: Total of all reporting groups
Arm/Group | Telerehabilitation - Infants | Home-based - Infants | Telerehabilitation -Mothers | Home-based - Mothers | Total
Number analyzed (Participants) | 13 | 13 | 13 | 13 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 0.54 (0.06) | 0.58 (0.07) | 28.85 (4.67) | 32.77 (5.29) | 15.68 (2.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13 | 13 | 39
  Male | 7 | 6 | 0 | 0 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Bayley III - Cognitive
Description: Cognitive development of infants will be evaluated.
  Standard Scores: The Cognitive Scale produces standard scores with a mean of 100 and a standard deviation of 15. Scores are typically categorized as follows:
  Above Average: >115 Average: 85-115 Below Average: <85 T-Scores: T-scores, commonly used in research, are derived with a mean of 50 and a standard deviation of 10. These scores are useful for comparing an individual's performance to normative data.
  Minimum and Maximum Scores:
  The floor score for the Cognitive domain in Bayley-III is 55, while the ceiling score is 145. These scores represent extreme levels of performance relative to the normative sample.
  Higher or Lower Scores:
  Higher Scores: Indicate better cognitive functioning or developmental progress. Lower Scores: Suggest potential delays or impairments in cognitive development.
Time Frame: Day 0
Population: Risky babies
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Telerehabilitation: A telerehabilitation-based exercise group where the therapist coaches the family, performs one-on-one exercises with families with a doll in his hand, and can perform the necessary interventions such as promoting good practices and preventing bad practices, and the other 2 days where the families show their exercises by sending videos to the therapist, and again provide the therapist's intervention and follow-up via videos
  Telerehabilitation: Family-centered, goal-oriented early physiotherapy approaches will be applied.
- Home-based: The Home-based group that will be given exercise training at the beginning of treatment and at 4., 8., and 12. week.
  Home-based: Family-centered, goal-oriented early physiotherapy approaches will be applied.
Arm/Group | Telerehabilitation | Home-based
Number analyzed (Participants) | 13 | 13
score on a scale | 77.69 (15.22) | 78.46 (14.19)

2. Primary Outcome: Bayley III - Cognitive Value at Day 30
Description: as for outcome 1
Time Frame: Day 30
Population: Risky babies
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telerehabilitation | Home-based
Number analyzed (Participants) | 12 | 12
score on a scale | 82.08 (11.76) | 77.08 (10.10)

3. Primary Outcome: Bayley III - Cognitive Value at Day 60
Description: as for outcome 1
Time Frame: Day 60
Population: Risky babies
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telerehabilitation | Home-based
Number analyzed (Participants) | 12 | 12
score on a scale | 84.58 (10.32) | 73.33 (12.67)

4. Primary Outcome: Bayley III - Cognitive Value at Day 90
Description: as for outcome 1
Time Frame: Day 90
Population: Risky babies
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telerehabilitation | Home-based
Number analyzed (Participants) | 12 | 12
score on a scale | 89.17 (7.63) | 82.08 (8.64)

5. Primary Outcome: Bayley III - Language
Description: Receptive Language: Measures how well a child understands spoken language and can respond to it.
  Expressive Language: Measures a child's ability to use words and sentences to communicate.
  Standard Scores: Like the Cognitive Scale, the Language subscale uses a mean of 100 and a standard deviation of 15. A typical distribution includes:
  Above Average: Scores above 115 Average: Scores between 85 and 115 Below Average: Scores below 85 The minimum score on the Bayley-III Language scale is 55, while the maximum is 145.
  Higher Scores: Indicate better language development and a stronger ability to understand and express language.
  Lower Scores: Suggest potential delays in language development, which may require further evaluation or intervention.
  T-Scores:
  The T-score for the Bayley-III Language scale is often used in research settings to compare an individual's performance against a larger population. Like standard scores, the mean is 50 and the standard deviation is 10.
Time Frame: Day 0
Population: Risky babies
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telerehabilitation | Home-based
Number analyzed (Participants) | 13 | 13
score on a scale | 77.85 (10.76) | 83.38 (7.27)

6. Primary Outcome: Bayley III - Language Value at Day 30
Description: as for outcome 5
Time Frame: Day 30
Population: Risky babies
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telerehabilitation | Home-based
Number analyzed (Participants) | 12 | 12
score on a scale | 85.17 (7.86) | 85.42 (4.92)

7. Primary Outcome: Bayley III - Language Value at Day 60
Description: as for outcome 5
Time Frame: Day 60
Population: Risky babies
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telerehabilitation | Home-based
Number analyzed (Participants) | 12 | 12
score on a scale | 84.83 (5.25) | 82.75 (4.39)

8. Primary Outcome: Bayley III - Language Value at Day 90
Description: as for outcome 5
Time Frame: Day 90
Population: Risky babies
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telerehabilitation | Home-based
Number analyzed (Participants) | 12 | 12
score on a scale | 89.92 (2.81) | 87.00 (5.76)

9. Primary Outcome: Bayley III - Motor
Description: Gross Motor: Assesses abilities related to large muscle groups. Fine Motor: Measures small muscle control. Standard Scores: The motor scale uses a mean of 100 and a standard deviation of 15, consistent with the Cognitive and Language scales.
  Above Average: Scores above 115. Average: Scores between 85 and 115. Below Average: Scores below 85. The minimum score on the Bayley-III Motor scale is 55, while the maximum is 145.
  T-Scores:
  The T-score is calculated using a mean of 50 and a standard deviation of 10, commonly used in research to compare an individual's performance with a larger population.
  Higher Scores: Indicate more advanced motor development, with better coordination and movement abilities.
  Lower Scores: Suggest potential delays in motor development, which may require intervention or further assessment.
Time Frame: Day 0
Population: Risky babies
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telerehabilitation | Home-based
Number analyzed (Participants) | 13 | 13
score on a scale | 81.08 (13.49) | 88.54 (11.14)

10. Primary Outcome: Bayley III - Motor Value at Day 30
Description: as for outcome 9
Time Frame: Day 30
Population: Risky babies
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telerehabilitation | Home-based
Number analyzed (Participants) | 12 | 12
score on a scale | 92.33 (12.07) | 88.08 (9.99)

11. Primary Outcome: Bayley III - Motor Value at Day 60
Description: as for outcome 9
Time Frame: Day 60
Population: Risky babies
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telerehabilitation | Home-based
Number analyzed (Participants) | 12 | 12
score on a scale | 89.00 (9.42) | 81.50 (8.93)

12. Primary Outcome: Bayley III - Motor Value at Day 90
Description: as for outcome 9
Time Frame: Day 90
Population: Risky babies
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telerehabilitation | Home-based
Number analyzed (Participants) | 12 | 12
score on a scale | 101.33 (5.86) | 95.08 (6.72)

13. Primary Outcome: Hammersmith Infant Neurological Examination (HINE)
Description: The total score is then calculated by summing the scores for all the items. A higher total score indicates more typical neurological development, while a lower score may indicate delays or neurological abnormalities.
  The HINE is divided in 3 sections. Section 1 (neurologic examination) consists of 26 items assessing cranial nerve function, posture, movements, tone, and reflexes and reactions, and the items are scored 0-3 points in 0.5-point steps with a maximum total score of 78.
  Interpretation:
  Normal: A total score of ≥57 generally indicates normal neurological function. Mild Abnormalities: Scores 46-56 suggest mild motor or neurological delays. Severe Abnormalities: Scores <45 are indicative of significant neurological concerns.
Time Frame: Day 0
Population: risky babies
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telerehabilitation | Home-based
Number analyzed (Participants) | 13 | 13
score on a scale | 51.92 (7.22) | 50.15 (7.09)

14. Primary Outcome: HINE Value at Day 30
Description: as for outcome 13
Time Frame: Day 30
Population: risky babies
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telerehabilitation | Home-based
Number analyzed (Participants) | 12 | 12
score on a scale | 58.08 (7.09) | 55.50 (6.08)

15. Primary Outcome: HINE Value at Day 60
Description: as for outcome 13
Time Frame: Day 60
Population: risky babies
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telerehabilitation | Home-based
Number analyzed (Participants) | 12 | 12
score on a scale | 66.50 (4.60) | 61.92 (6.14)

16. Primary Outcome: HINE Value at Day 90
Description: as for outcome 13
Time Frame: Day 90
Population: risky babies
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telerehabilitation | Home-based
Number analyzed (Participants) | 12 | 12
score on a scale | 74.00 (3.24) | 68.92 (6.59)

17. Primary Outcome: Goal Attainment Scale (GAS)
Description: Goal Attainment Scaling (GAS) allows clinicians or educators to establish specific, individualized goals for a patient or student. These goals are tailored to the individual's needs and context and are evaluated using a 5-point ordinal scale that includes both positive and negative values:
  The 5-point scale includes:
  "plus two" (much better than expected), "plus one" (slightly better than expected), "zero" (expected outcome), "minus one" (slightly worse than expected), and "minus two" (much worse than expected).
Time Frame: Day 0
Population: risky babies
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telerehabilitation | Home-based
Number analyzed (Participants) | 13 | 13
score on a scale | -1.62 (0.76) | -0.85 (1.06)

18. Primary Outcome: GAS Value at Day 30
Description: as for outcome 17
Time Frame: Day 30
Population: risky babies
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telerehabilitation | Home-based
Number analyzed (Participants) | 12 | 12
score on a scale | -0.42 (1.37) | -1.25 (0.96)

19. Primary Outcome: GAS Value at Day 60
Description: as for outcome 17
Time Frame: Day 60
Population: risky babies
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telerehabilitation | Home-based
Number analyzed (Participants) | 12 | 12
score on a scale | -0.33 (0.88) | -1.25 (0.75)

20. Primary Outcome: GAS Value at Day 90
Description: as for outcome 17
Time Frame: Day 90
Population: risky babies
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telerehabilitation | Home-based
Number analyzed (Participants) | 12 | 12
score on a scale | 0.50 (0.90) | -0.50 (0.67)

21. Other Pre Specified Outcome: Telerehabilitation Satisfication Survey
Description: This questionnaire was developed by the researchers to assess parental satisfaction with the telerehabilitation process. It includes 8 items focusing on perceived effectiveness, convenience, communication quality, and technical usability of the sessions.
  Scale: Each item is rated on a 5-point Likert scale ranging from 1 (Strongly Disagree) to 5 (Strongly Agree).
  Total Score Range: 8 (minimum satisfaction) to 40 (maximum satisfaction). Scoring: The total satisfaction score is obtained by summing the scores of all 8 items. Higher scores indicate greater satisfaction with the telerehabilitation experience. There are no subscales and no reverse-scored items.
Time Frame: Day 90
Population: Mothers of risky babies
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Telerehabilitation | Home-based
Number analyzed (Participants) | 12 | 12
score on a scale | 40 [38.25 to 40] | 35.5 [35 to 36]

ADVERSE EVENTS:
Time Frame: Measured at 12 weeks post-baseline (Week 12 of intervention.)
Groups:
- Home-based: The home-based group that will be given exercise training at the beginning of treatment and at 4., 8., and 12.
  Home-based: Family-centered, goal-oriented early physiotherapy approaches will be applied.
Arm/Group | Telerehabilitation | Home-based
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-02): https://cdn.clinicaltrials.gov/large-docs/24/NCT05333224/Prot_SAP_000.pdf